CLINICAL TRIAL: NCT07253051
Title: BRCA Mutation Carriers' Platform, a Multicenter Study
Brief Title: BRCA Mutation Carriers' Platform a Multicenter Study
Acronym: BRCA_ENDORSE
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4224
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: BRCA1 Mutation; BRCA2 Mutation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Registration of clinical datas in the platform — Registration of clinical datas in the platform of female individual carrying a BRCA1 or BRCA2 mutation

SUMMARY:
Subjects who carry mutations in breast cancer susceptibility genes 1 and 2 (BRCA1 and BRCA2 genes) are at higher risk of developing cancers. Despite the cumulative amount of evidence published in the literature in the last two decades, the management of BRCA mutation carriers is still not completely defined.

Since the prevalence of the mutation is estimated to be 1:400 - 1:500 individuals, the total number of BRCA mutation carriers should be around 140.000 - 150.000 in the Italian population. It is estimated that 87% of women with BRCA mutations will experience, in their lifetime, a tumor with a genetic origin. About 20% of the 5200 ovarian cancer cases diagnosed each year in Italy has a genetic origin and could potentially be the object of primary prevention. To date, and to the best of our knowledge, a national prospective data collection on women with BRCA mutations has not been yet established.

ELIGIBILITY:
Inclusion Criteria:

* All women who are 18 years of age or older;
* All women who known to be carriers of a pathogenetic mutation class 4 and 5 of the International Agency of Research on Cancer classification) of the BRCA1 or BRCA2 genes.

Exclusion Criteria:

* Age < 18 years old;
* No pathogenetic mutation carriers.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women who are 18 years of age or older and known to be carriers of a pathogenetic mutation class 4 and 5 of the International Agency of Research on Cancer classification) of the BRCA1 or BRCA2 genes, who signed Informed Consent.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-04-05 (Actual); Primary Completion 2045-04-01 (Estimated); Study Completion 2045-12-31 (Estimated)

PRIMARY OUTCOMES:
Collection data about BRCA mutation | 1 day
  To collect data of each female individual carrying a BRCA1 or BRCA2 mutation

SECONDARY OUTCOMES:
GEOGRAPHICAL DISTRIBUTION OF BRCA MUTATIONS | 6 months
  GEOGRAPHICAL DISTRIBUTION OF BRCA MUTATIONS FOR IDENTIFY THE AREAS WHERE THE INCIDENCE OF THE MUTATION IS HIGHER THAN EXPECTED
CENTRALIZATION OF CASES IN HIGHLY SPECIALIZED CENTERS | 6 months
  CENTRALIZATION OF CASES IN HIGHLY SPECIALIZED CENTERS FOR THE PREVENTION AND TREATMENT OF GENETIC-RELATED CANCER
RELATIONSHIP BETWEEN SPECIFIC MUTATIONS AND SPECIFIC TYPES OF CANCER | 6 months
  DEFINITION OF THE RELATIONSHIP BETWEEN SPECIFIC MUTATIONS AND THE ONSET OF SPECIFIC TYPES OF CANCER
CRITERIA FOR DETERMINING THE ACCESS TO GENETIC EVALUATION | 6 months
  EVALUATION OF THE ADEQUACY OF THE CRITERIA FOR DETERMINING THE ACCESS TO GENETIC EVALUATION
LIFESTYLE RISK FACTORS | 6 months
  DEFINITION OF LIFESTYLE RISK FACTORS FOR THE DEVELOPMENT OF TUMORS IN BRCA MUTATION CARRIERS
DEFINITION OF PREVENTIVE STRATEGIES | 6 months
  HEALTHY SUBJECTS: DEFINITION OF RISK REDUCING OR PREVENTIVE STRATEGIES
Risk-reducing salpingo-oophorectomy | 6 months
  MANAGEMENT OF WOMEN AFTER RRSO (risk-reducing salpingo-oophorectomy) AFTER SURGERY

CONTACTS AND LOCATIONS:
Overall Officials: Anna Fagotti, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (39):
- Italy (39):
  - Malzoni Research Hospital, Avellino
  - Centro di Riferimento Oncologico IRCCS, Aviano
  - Università degli Studi di Bari "Aldo Moro", Bari
  - IRCCS Istituto Tumori "Giovanni Paolo II", Bari
  - ASST Papa Giovanni XXIII, Bergamo
  - L'Azienda ospedaliera per l'emergenza "Cannizzaro", Catania
  - Azienda Ospedaliero Santa Croce e Carle, Cuneo
  - Presidio Ospedaliero Umberto I - ASP di Enna, Enna
  - Azienda Ospedaliero Universitaria Careggi, Oncologia Medica Ginecologica, Florence
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Ospedale S. Maria Goretti, Latina, Latina
  - Ospedale del Tigullio Polo di Lavagna - ASL 4 Chiavarese, Lavagna
  - Ospedale Vito Fazzi, Lecce, Lecce
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori", Meldola
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Humanitas San Pio X - Milano, Milan
  - Presidio Ospedaliero di Mirano, Mirano
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - Ospedale Mater Olbia, Olbia
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliera Universitaria di Parma, Parma
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Centro Nazionale di Adroterapia Oncologica, Pavia
  - Fondazione I.R.C.C.S. Policlinico San Matteo, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Policlinico Umberto I Università "La Sapienza", Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, UOC Ginecologia Oncologica, Rome
  - Azienda Ospedaliera Universitaria Senese, Siena
  - Ospedale G. Mazzini di Teramo, Teramo
  - Azienda sanitaria universitaria Friuli Centrale, Tolmezzo
  - Azienda Ospedaliero Universitaria Citta della Salute e della Scienza di Torino, Torino
  - Ospedale Mauriziano Umberto I, Torino
  - Azienda ULSS 2 MARCA TREVIGIANA, Treviso
  - IRCCS materno infantile Burlo Garofolo, Trieste
  - Azienda Ospedaliera Universitaria Integrata, Verona
  - AULSS 8 Berica, Vicenza